CLINICAL TRIAL: NCT04224675
Title: Captopril Versus Atenolol to Prevent Expansion Rate of Thoracic Aortic Aneurysms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Onassis Cardiac Surgery Centre (Other)
Responsible Party: Principal Investigator, Michael Spartalis, MD, MSc, FESC, FEHRA, FACC, CCDS, Onassis Cardiac Surgery Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OnassisCSC
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Aneurysm
MeSH Terms: conditions — Aneurysm | interventions — Atenolol; Captopril

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ate (Other)
  Interventions: Drug: Atenolol
- Cap (Other)
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Atenolol — Captopril versus atenolol to prevent expansion rate of thoracic aortic aneurysms
  Other Names: Captopril

SUMMARY:
Thoracic aortic aneurysms (TAA) are considered "silent killers" because they scarcely display any symptomatology, but are correlated with significant mortality and morbidity. Current guidelines regard aortic aneurysm disease as a coronary artery disease equivalent and suggest aspirin and statin use to reduce the progression of atherosclerosis, as well as beta-blocker (BB) therapy. No therapy, however, is effective at limiting aneurysm expansion and preventing rupture, even in large trials. TAA has emerged as an inflammation-mediated disorder. Angiotensin-converting enzyme inhibitors (ACEIs) can reduce the wall shear stress and inflammation, both of which play vital roles in the expansion of the aneurysm.

The study will be a randomized, double-blind trial. Patients will be randomized into one of two parallel arms, receiving captopril or atenolol. The doses of captopril and atenolol will be 25 mg daily for the first 15 days, rising to 100 mg according to clinical tolerance and BP estimates. The sample size will be set at 424 subjects (212 per group). The primary end-point will be the rate of change in the absolute diameter of the aortic root and ascending aorta on MRI of the aorta after 36 months of therapy with captopril vs. atenolol.

BBs have not been precisely found to decrease aneurysm growth rates. ACEIs could lead to the prevention of aneurysm degeneration through their antihypertensive and anti-inflammatory properties.

The results of this trial will clarify that ACEIs are superior to BB therapy in reducing the growth rate of TAAs, the rate of change in aortic insufficiency, the time to aortic rupture or dissection, the need for aortic surgery or intervention, and death.

ELIGIBILITY:
Inclusion Criteria:

All adult men or women, aged at least 70 years, with TAA 3.0-5.5 cm in diameter measurements according to magnetic resonance imaging (MRI) of the aorta and with a systolic BP < 150 mmHg will be eligible for inclusion in the study.

Exclusion Criteria:

Patients already receiving an ACEI or BB daily, patients with known renal artery stenosis (> 50%), patients incapable of providing informed consent, history of aortic dissection, angioedema or any intolerance to ACEIs or BBs, asthma, pregnancy, frailty, respiratory failure, and renal failure.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2020-03-07 (Estimated); Primary Completion 2023-03-07 (Estimated); Study Completion 2023-03-07 (Estimated)

PRIMARY OUTCOMES:
rate of change in the absolute diameter of the aortic root and ascending aorta on MRI of the aorta after 36 months of therapy with captopril vs. atenolol | 3 years

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Spartalis M, Tzatzaki E, Iliopoulos DC, Spartalis E, Patelis N, Athanasiou A, Paschou SA, Voudris V, Siasos G. Captopril versus atenolol to prevent expansion rate of thoracic aortic aneurysms: rationale and design. Future Cardiol. 2021 Mar;17(2):189-195. doi: 10.2217/fca-2020-0062. Epub 2020 Aug 25. PMID 32842783